CLINICAL TRIAL: NCT04725851
Title: High Concentration of Inspired Oxygen for Pneumocephalus After Evacuation of Chronic Subdural Haematoma: A Randomized Controlled Trial (HOPE Study)
Brief Title: High Concentration Oxygen for Pneumocephalus After Evacuation of Chronic Subdural Haematoma
Acronym: HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. David Yuen Chung CHAN, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2021-0021
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Chronic Subdural Hematoma; Recurrence; Oxycephaly
Keywords: Chronic subdural hematoma; Oxygen therapy; Normobaric Oxygen; High concentration Oxygen; Pneumocephalus; Recurrence
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence; Craniosynostoses; Pneumocephalus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High concentration Oxygen Therapy (Experimental): 12-15 Litre/min O2 delivery via Non-Rebreather Mask (NRM) consecutively for 24 hours.
  Interventions: Procedure: High concentration Oxygen therapy
- Room air or low concentration oxygen (Placebo Comparator): Room air or low concentration oxygen (0-2 Litre/min O2 ) consecutively for 24 hours.
  Interventions: Procedure: Control: Room Air or Low concentration Oxygen

INTERVENTIONS:
Procedure: High concentration Oxygen therapy — FiO2 >80% Oxygen (Delivered with 12-15L/min Non-rebreather Mask)
  Arms: High concentration Oxygen Therapy
Procedure: Control: Room Air or Low concentration Oxygen — FiO2 <30% Oxygen (Delivered with 0-2L/min Nasal Cannula)
  Arms: Room air or low concentration oxygen

SUMMARY:
Normobaric oxygen therapy was shown to be effective in reducing post craniotomy pneumocephalus. Theoretical assessment of normobaric oxygen therapy in treating pneumocephalus has shown that a higher level of oxygen concentration will significantly decrease the time for absorption of pneumocephalus. The therapeutic efficacy is not fully established in patients with chronic subdural hematoma after burr hole drainage. Both radiological outcomes and clinical outcomes would be evaluated.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is not a benign disease. Morbidity and mortalities were high especially in those with recurrence requiring reoperations. The use of subdural drain after burr hole drainage is an excellent example demonstrating that by reducing CSDH recurrence, a significant improvement in functional outcomes can be observed.

Pneumocephalus is very common after burr hole drainage for CSDH. The use of high-flow oxygen had been reported to be effective in small case series, showing effectiveness in clinical and radiological outcomes. However, no large, prospective, controlled trial has been conducted to establish the efficacy of oxygen therapy on functional outcomes for patients with pneumocephalus after burr hole drainage in CSDH.

Bilateral CSDH has a different prognosis and is associated with a poorer outcome.

In addition to treating pneumocephalus, the use of perioperative oxygen has been suggested to minimize tissue hypoxemia and infection. In a study published in the New England Journal of Medicine, the use of perioperative supplementary oxygen was shown to reduce surgical site infection.

Hyperoxia with oxygen therapy has shown to be safe with minimal changes to the cerebral blood flow (CBF) from functional magnetic resonance imaging (fMRI).

Research Questions

1. Does post-operative high-flow oxygen improve pneumocephalus in terms of volume reduction in CSDH patients after burr-hole drainage?
2. Does post-operative high-flow oxygen reduce the recurrence rate of CSDH (radiologically) if pneumocephalus volume is reduced after oxygen therapy?
3. Does post-operative high-flow oxygen reduce the recurrence rate of CSDH (clinically), as defined by symptomatic recurrence requiring reoperation, if pneumocephalus volume is reduced after oxygen therapy?
4. Does post-operative high-flow oxygen improve CSDH patients' functional outcome in terms of modified Rankin Scale (mRS) at 3 months and 6 months?

Hypothesis Oxygen therapy for CSDH patients with post-operative pneumocephalus will experience significant resorption of intracranial air within 24 hours. There is a reduction in recurrence rate in terms of the re-operation rates. There is an improvement in functional outcome in terms of mRS.

Aim of the Study To evaluate changes in pneumocephalus volume and functional outcome after oxygen therapy in post-operative CSDH patients treated by burr hole drainage, as compared to the standard care by breathing in room air or low concentration oxygen during the post-operative period.

Study Design Prospective randomized 1:1 parallel-arm study

Methods and Randomization Patients will be recruited when they are considered fit for oxygen therapy as determined by the treating clinician. The timing of burr hole evacuation may vary according to the availability of the emergency operative time slot. The index intervention is postoperative oxygen therapy: 100% normobaric oxygen through a nonrebreather mask (NRM) at 12-15 Litre/minute consecutively for 24 hours. Removal of the nonrebreather mask is allowed during meals or other activities such as physiotherapy. The duration of mask removal would be documented. Compliance with NRM is considered to be good if the mask is kept > 90% of the time during the 24 hours treatment period. The reference intervention is standard post-operative care: the patient would be breathing in normobaric room air. For the reference arm, if the patient has desaturation (i.e. SaO2 < 93%), supplemental O2 therapy can be given to keep SaO2 > 93%. Arterial blood gas would be obtained by the clinicians when deemed necessary. If there is a significant deviation from the study protocol occurs, the patients will be analyzed according to their originally assigned groups (intention-to-treat principle).

Non-rebreather masks, when they are tightly applied, are associated with a lower aerosol dispersion distance (as compared to non-invasive positive pressure ventilation or venturi masks).

Interim data analysis would be performed and the study would be terminated if a significant difference in the primary outcome is observed.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years-old.
2. Presence of chronic subdural haematoma (CSDH) as diagnosed radiologically either by computed tomography (CT) brain scan or magnetic resonance imaging (MRI).
3. Treatment of CSDH by burr-hole evacuation.
4. Presence of post-operative pneumocephalus, as evidenced from post-operative CT Brain or MRI brain
5. Negative test to SARS-nCoV-2, as evidenced by either deep throat saliva rapid test, deep throat saliva PCR test, nasopharyngeal swab real-time PCR test, or nasopharyngeal swab rapid test within seven days.

Exclusion Criteria:

1. Presence of pre-existing respiratory conditions such as chronic obstructive pulmonary disease (COPD) and hence not suitable for oxygen therapy.
2. Any pre-existing illness that renders the patient moderately or severely disabled before diagnosis with CSDH, such as a history of central nervous system infection.
3. CSDH arising from secondary causes, such as intracranial hypotension, thrombocytopenia, etc.
4. Any evidence or suspicion that there is communication between the pneumocephalus with the air cells (e.g. such as mastoid air cells) or air sinuses (e.g. frontal sinus).
5. Patients that need an additional procedure e.g. epidural blood patch, etc.
6. Complications arising from the burr-hole operation or subdural drain insertion such as hemorrhage or surgical site infection requiring surgical intervention or deemed to affect the patient's long-term functional outcome.
7. Patients already on long-term steroid for pre-existing medical conditions.
8. Participation in other clinical trials within four weeks upon recruitment.
9. Pregnancy or on breastfeeding.
10. Any other reasons that the researchers consider the patients to be unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the volume of pneumocephalus after 24 hours of oxygen therapy | 24 hours
  Volumetric measurement of pneumocephalus from Computed Tomographic (CT) scan for the Head

SECONDARY OUTCOMES:
Modified Rankins Scale (mRS) | at baseline before admission, on admission, at 1 month, at 3 months and at 6 months.
  Functional outcomes
EuroQOL EQ-5D | at 1 month, at 3 months and at 6 months.
  Functional outcomes
Glasgow Coma Scale (GCS) | On admission, at 1 month, at 3 months and at 6 months.
  Neurological examination
Recurrence rate, as defined by reoperation rate due to symptomatic recurrence | Reoperation rate within six months, including the number of re-operations for CSDH during the same admission episode, as well as subsequent readmission for reoperation for CSDH.
  Surgical complications
Changes in brain volume re-expansion | after 24 hours of oxygen therapy and 1 week after oxygen therapy
  Volumetric measurement from Computed Tomographic (CT) scan for the Head
Changes in volume of subdural fluid | Recurrence or re-accumulation rate, as measured by an increase in subdural fluid volume at 1 week, 1 month, 3 months, and at 6 months.
  Volumetric measurement from Computed Tomographic (CT) scan for the Head
Incidence of superficial wound infection | Any surgically associated would infections within 6 months from the index operation
  Surgical complications
Incidence of deep wound infection, including subdural empyema | Any surgically associated would infections within 6 months from the index operation
  Surgical complications
Incidence of chest complications, including chest infection | Any complications within the same admission episode for the index operation
  Complications
Any complications arising from the Oxygen therapy (Adverse events) | Any complications within the same admission episode for the index operation
  Complications
Barthel Index | at 1 month, 3 months and 6 months
  Functional outcome
PaO2 and PaCO2 from the arterial blood gas (ABG) | During oxygen therapy
  Blood taking for ABG when judged to be necessary by the treating physician or when there is desaturation to SaO2 < 93%
Duration of stay at the acute neurosurgical ward (LOS) | During the same admission episode for the index operation
  LOS
Discharge destination | Upon the same admission episode for the index operation
  Outcome
The length of stay in secondary care | Upon transferal to the secondary care from the same admission episode for the index operation
  LOS
Mortality rate at 30 days, 3 months and 6 months. | at 30 days, 3 months and 6 months.
  Death rate

OTHER OUTCOMES:
Recurrence rate in BILATERAL Chronic Subdural Hematoma (CSDH) | Within six months from the index operation
  Bilateral (CSDH)
Volumetric reduction in pneumocephalus in BILATERAL Chronic Subdural Hematoma (CSDH) after Oxygen therapy | Within 24 hours after Oxygen therapy
  Bilateral (CSDH)
Improvement in mRS for BILATERAL Chronic Subdural Hematoma (CSDH) | at 1 month, 3 months and 6 months
  Functional outcome in bilateral CSDH

CONTACTS AND LOCATIONS:
Overall Officials: David YC Chan, MBBS, FRCS, Principal Investigator — Chinese University of Hong Kong; Wai S Poon, MBChB, FRCS, Study Chair — Chinese University of Hong Kong
Locations (1):
- Division of Neurosurgery, Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gore PA, Maan H, Chang S, Pitt AM, Spetzler RF, Nakaji P. Normobaric oxygen therapy strategies in the treatment of postcraniotomy pneumocephalus. J Neurosurg. 2008 May;108(5):926-9. doi: 10.3171/JNS/2008/108/5/0926. PMID 18447708
- [Background] Dexter F, Reasoner DK. Theoretical assessment of normobaric oxygen therapy to treat pneumocephalus. Anesthesiology. 1996 Feb;84(2):442-7. doi: 10.1097/00000542-199602000-00024. PMID 8602677
- [Background] Greif R, Akca O, Horn EP, Kurz A, Sessler DI; Outcomes Research Group. Supplemental perioperative oxygen to reduce the incidence of surgical-wound infection. N Engl J Med. 2000 Jan 20;342(3):161-7. doi: 10.1056/NEJM200001203420303. PMID 10639541
- [Background] Xu F, Liu P, Pascual JM, Xiao G, Lu H. Effect of hypoxia and hyperoxia on cerebral blood flow, blood oxygenation, and oxidative metabolism. J Cereb Blood Flow Metab. 2012 Oct;32(10):1909-18. doi: 10.1038/jcbfm.2012.93. Epub 2012 Jun 27. PMID 22739621
- [Background] Santarius T, Kirkpatrick PJ, Ganesan D, Chia HL, Jalloh I, Smielewski P, Richards HK, Marcus H, Parker RA, Price SJ, Kirollos RW, Pickard JD, Hutchinson PJ. Use of drains versus no drains after burr-hole evacuation of chronic subdural haematoma: a randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1067-73. doi: 10.1016/S0140-6736(09)61115-6. PMID 19782872
- [Background] Miranda LB, Braxton E, Hobbs J, Quigley MR. Chronic subdural hematoma in the elderly: not a benign disease. J Neurosurg. 2011 Jan;114(1):72-6. doi: 10.3171/2010.8.JNS10298. Epub 2010 Sep 24. PMID 20868215
- [Background] Chan DYC, Poon WS, Chan DTM, Mak WK, Wong GKC. Chronic subdural haematoma during the COVID-19 lockdown period: late presentation with a longer interval from the initial head injury to the final presentation and diagnosis. Chin Neurosurg J. 2021 Jan 8;7(1):4. doi: 10.1186/s41016-020-00229-7. PMID 33419483
- [Background] Chan DY, Woo PY, Mak CH, Chu AC, Li CC, Ko NM, Ng SC, Sun TF, Poon WS. Use of subdural drain for chronic subdural haematoma? A 4-year multi-centre observational study of 302 cases. J Clin Neurosci. 2017 Feb;36:27-30. doi: 10.1016/j.jocn.2016.10.039. Epub 2016 Nov 30. PMID 27914805
- [Background] Chan DY, Chan DT, Sun TF, Ng SC, Wong GK, Poon WS. The use of atorvastatin for chronic subdural haematoma: a retrospective cohort comparison study. Br J Neurosurg. 2017 Feb;31(1):72-77. doi: 10.1080/02688697.2016.1208806. Epub 2016 Nov 23. PMID 27881024
- [Background] Chan DYC, Sun TFD, Poon WS. Steroid for chronic subdural hematoma? A prospective phase IIB pilot randomized controlled trial on the use of dexamethasone with surgical drainage for the reduction of recurrence with reoperation. Chinese Neurosurgical Journal. 2015; 1(1):2.